CLINICAL TRIAL: NCT02398968
Title: Effect of Iron Supplementation on Recurrent Upper Respiratory Tract Infections in Egyptian School Children: A One Year Prospective Study
Brief Title: Iron Supplementation Outcome on Recurrent Upper Respiratory Tract Infections in 6-15 Years Old Egyptian School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, yasmin gamal el gendy, lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-elalfy
Record Dates: First submitted 2015-02-19; First posted 2015-03-26 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Upper Respiratory Tract Infections; Iron Deficiency Anemia
Keywords: Iron; RURTIs; CARIFS; children
MeSH Terms: conditions — Respiratory Tract Infections; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RURTI+IDA+iron therapy (Active Comparator): children with iron deficiency anemia on therapeutic iron fumerate therapy (6mg/kg/d) for 3 months, then maintained on iron fumerate supplementation(1mg/kg/d) for 12 months
  Interventions: Dietary Supplement: iron fumerate
- B1:RURTI+no anemia+iron maintenance (Active Comparator): children with recurrent upper respiratory tract infection and no anemia receiving oral iron fumerate (1mg/kg/d) for 12 months
  Interventions: Dietary Supplement: iron fumerate
- B2:RURTI+no anemia (No Intervention): children with recurrent upper respiratory tract infection and no anemia followed up for 12 months

INTERVENTIONS:
Dietary Supplement: iron fumerate — iron fumerate supplementation (6mg/kg/d) for arm 1 iron fumerate supplementation (1mg/kg/d) for arm 2
  Arms: B1:RURTI+no anemia+iron maintenance; RURTI+IDA+iron therapy

SUMMARY:
Recurrent upper respiratory infections ( RURTIs) are common in school aged children. An adequate iron status might reduce their prevalence. The aim of the study is to assess the percentage and type of RURTIs in Egyptian school children, assessing the percentage of iron deficiency anemia (IDA) and the effect of iron supplementation on the recurrence and severity of upper respiratory tract infections .

DETAILED DESCRIPTION:
This is a prospective interventional study in which 1000 Children (6-15 years) are recruited from two schools in urban Cairo; three months enrollment was done in early autumn ; students defined to have RURTIs were screened by Hemocue; if anemic (Hb < 11.5gm/dL),Complete blood picture and iron profile were done, they were enrolled into 2 groups: (A)children with IDA on oral iron fumerate therapy (6mg/kg/d) for 3 months, then maintained on oral iron (1mg/kg/d) for 12 months, and (B) Non anemic group; were randomly assigned in 1:1 ratio into: group (B1)children Received maintenance iron therapy for 12 months and group (B2) received placebo. Recurrence and severity of URTIs using (CARIFS score) throughout the study are recorded

ELIGIBILITY:
Inclusion Criteria:

* Both genders were eligible, and we did not seek to balance the number of boys and girls.
* Children completed the compulsory vaccination schedule of Egypt.

Exclusion Criteria:

* Children with coexisting chronic disease such as renal, hepatic failure , IDDM, endocrine diseases, bronchial asthma and chronic diarrhea .
* Patients with suspected immunodeficiency by presence of some of the warning symptoms or signs .

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
effect of iron supplementation on recurrent upper respiratory tract infections measured by Canadian Acute Respiratory Illness and Flu Scale {CARIFS} | 15 months
  Assessment of the upper respiratory tract infection incidence and severity throughout the study period will be done by a questionnaire including: Number of upper respiratory tract infection episodes per month with or without absenteeism from school, Total number of days sick with an upper respiratory tract infection ,and Canadian Acute Respiratory Illness and Flu Scale {CARIFS}

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, professor, Study Director — Ain Shams University; Ehab K Emam, professor, Study Chair — Ain Shams University; Khaled M Abd-al aziz, professor, Study Chair — Ain Shams University; Yasmin G El gendy, lecturer, Principal Investigator — Ain Shams University; Mohamed T Hamza, lecturer, Study Chair — Ain Shams University; marian g rizk, ass lect, Principal Investigator — Ain Shams University
Locations (1):
- Pediatrics hospital Ain shams University, Cairo, Egypt